CLINICAL TRIAL: NCT00627055
Title: The HIV Second-line Therapy AntiRetroviral Study in Patients Who Failed NNRTI-based Regimens
Brief Title: Second-line Therapy Antiretroviral in Patients Who Failed Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) - Based Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: National Health Security Office, Thailand (Other); Swiss HIV Cohort Study (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 079; IRB#417/70
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Second line antiretroviral therapy; HIV genotypic resistance; Kaletra monotherapy; Thailand; 48-week efficacy and safety between 2 NRTIs plus lopinavir/ritonavir (LPV/r) and LPV/r monotherapy in patients failing a standard NNRTI-based treatment regimen; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): LPV/r monotherapy
  Interventions: Drug: LPV/r
- 2 (Active Comparator): LPV/r + 2NRTIs (TDF/FTC or TDF/3TC)
  Interventions: Drug: LPV/r + TDF/FTC or TDF/3TC

INTERVENTIONS:
Drug: LPV/r — LPV/r dosing = 400mg/100mg orally q12h for 48 weeks
  Arms: 1
Drug: LPV/r + TDF/FTC or TDF/3TC — TDF/FTC (Truvada) 1 pill orally q 24 hr or TDF 300mg orally q 24 hr/3TC 300mg orally q 24 hr (or 3TC 150mg orally q 12 hr) for 48 weeks
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety at 48 weeks between LPV/r monotherapy and 2 NRTIs + LPV/r therapy in patients failing a standard NNRTI-based treatment regimen. Also, to evaluate the short-term 24-week efficacy and safety of Lopinavir/ritonavir (LPV/r) monotherapy and 2 NRTIs+LPV/r therapy in patients failing a standard NNRTI-based treatment regimen as an interim analyses when 50% of the patients in each arm have reached 24 weeks after randomization. Last, to define risk factors for monotherapy failure in HIV-treated individuals

Hypothesis. The rate of virologic suppression is not inferior in the monotherapy arm.

DETAILED DESCRIPTION:
With at least 80,000 HIV-1 infected individuals throughout Thailand currently on generically produced fixed dose combination of d4T/3TC/NVP or GPOvir as a first line national recommendation therapy, we will inevitably face with resistance problem in a large number of patients near future. Therefore a comprehensive investigation into the best second line regimen for these individuals is needed. Given the situation in Thailand where economic burden is a major challenge, the second line regimen will have to offer the greatest possible efficacy, and cost-effectiveness.

Second-line therapies necessitate treatment with combinations of drugs including protease inhibitors[3]. Such high drug concentrations can be achieved by combining protease inhibitors (such as indinavir, saquinavir, amprenavir and lopinavir) with ritonavir (RTV), known to boost the other protease plasma levels through potent inhibition of the cytochrome P450. Low dose RTV (100mg bid) significantly improves pharmacokinetics (AUC and plasma half life) of most protease inhibitors with the exception of nelfinavir. However, these combinations are more expensive, particularly if NRTIs are continued. In addition to increasing cost, continuing NRTIs may not add to the antiviral effect (if resistance is present) and may prolong the toxicity observed during the previous regimen.

Mono boosted PI therapy trials in HIV adults, as maintenance therapy after suppressed viral load, have been shown to be effective and safe [4-6]. This strategy not only decreases number of pill per dose but also saves ARV cost and might improve patient's adherence.

Lopinavir/ritonavir (LPV/r) is widely used protease inhibitor because of its high efficacy and high genetic barrier. As maintenance monotherapy after HIV-1 viral suppression, LPV/r has shown efficacy in 4 adult trials with 81-94% virological suppression[4, 7]. In the OK study[4], the virological failure cases had significantly higher missed doses (p = 0.008). Viral re-suppression after reintroduction of 2NRTIs was achieved in the LPV/r monotherapy arm. A pilot study of switch to LPV/r monotherapy from NNRTI-based therapy was reported with 92% participants on treatment at week 48 having HIV RNA <75 copies/mL[8].

In the OK04 study[9], 196 patients were randomized to eitherLPV/r monotherapy or LPV/r plus 2NRTIs. The percentage of viral suppression to < 50 copies/ml, at week 96 was 77% in the LPV/r monotherapy arm and 78% in the LPV/r plus 2NRTIs arm.

In the MONARK study, LPV/r monotherapy was used in 138 naïve adults and the percentage of viral suppression at week 48 was 71% compared to 75% in the LPV/r plus AZT and 3TC arm[10] (p = 0.69). Two patients in LPV/r monotherapy developed PI mutations but both were able to resuppress HIV-RNA when NRTIs were added. Neither patient displayed phenotypic resistance to LPV/r.

Therefore, we propose this comprehensive study to guide us in identifying the best second line regimen in order to prepare for the large scale antiretroviral resistance problem in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* HIV seropositive.
* Have had NNRTI-based HAART in the past for at least 6 months
* Naïve to protease inhibitors (PIs)
* Plasma HIVRNA ≥ 1000 copies/ml
* Signed written informed consent

Exclusion Criteria:

* Active AIDS-defining disease or active opportunistic infection
* Previously treated with PIs
* Pregnancy (negative pregnancy test for women of childbearing potential at screening).
* Documented chronic hepatitis B (HbsAg positive)
* ALT ≥ 200 U/L
* Creatinine clearance < 60 c.c. per min by Cockroft-Gault formula formula
* Use of medication that interfere with the action of LPV/r

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the 48-week efficacy and safety between 2 NRTIs plus lopinavir/ritonavir (LPV/r) and LPV/r monotherapy in patients failing a standard NNRTI-based treatment regimen | 48 weeks

SECONDARY OUTCOMES:
To evaluate the short-term 24-week efficacy and safety of LPV/r monotherapy and interim analyses when 50% of the patients in each arm have reached 24 weeks after randomization 2. To define risk factors for monotherapy failure in HIV-treated individuals | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — HIV-NAT, The Thai Red Cross AIDS Research Centre (TRCARC), and Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand; Bernard Hirschel, MD, Principal Investigator — Geneva University, Geneva, Switzerland
Locations (10):
- Thailand (10):
  - Chonburi Hospital, Chon Buri, Changwat Chon Buri
  - Chulalongkorn University, Bangkok
  - Hivnat, Trcarc, Bangkok
  - Siriraj Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Taksin Hospital, Bangkok
  - Sanpatong Hospital, Chiang Mai
  - Chiang Rai Regional Hospital, Chiang Rai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi

REFERENCES:
- [Derived] Parsons MS, Madhavi V, Ana-Sosa-Batiz F, Center RJ, Wilson KM, Bunupuradah T, Ruxrungtham K, Kent SJ. Brief Report: Seminal Plasma Anti-HIV Antibodies Trigger Antibody-dependent Cellular Cytotoxicity: Implications for HIV Transmission. J Acquir Immune Defic Syndr. 2016 Jan 1;71(1):17-23. doi: 10.1097/QAI.0000000000000804. PMID 26761269
- [Derived] Bunupuradah T, Chetchotisakd P, Ananworanich J, Munsakul W, Jirajariyavej S, Kantipong P, Prasithsirikul W, Sungkanuparph S, Bowonwatanuwong C, Klinbuayaem V, Kerr SJ, Sophonphan J, Bhakeecheep S, Hirschel B, Ruxrungtham K; HIV STAR Study Group. A randomized comparison of second-line lopinavir/ritonavir monotherapy versus tenofovir/lamivudine/lopinavir/ritonavir in patients failing NNRTI regimens: the HIV STAR study. Antivir Ther. 2012;17(7):1351-61. doi: 10.3851/IMP2443. Epub 2012 Jul 2. PMID 23075703
- [Derived] Bunupuradah T, Chetchotisakd P, Jirajariyavej S, Valcour V, Bowonwattanuwong C, Munsakul W, Klinbuayaem V, Prasithsirikul W, Sophonphan J, Mahanontharit A, Hirschel B, Bhakeecheep S, Ruxrungtham K, Ananworanich J; HIV STAR Study Group. Neurocognitive impairment in patients randomized to second-line lopinavir/ritonavir-based antiretroviral therapy vs. lopinavir/ritonavir monotherapy. J Neurovirol. 2012 Dec;18(6):479-87. doi: 10.1007/s13365-012-0127-9. Epub 2012 Sep 20. PMID 22993101
- [Derived] Bunupuradah T, Ananworanich J, Chetchotisakd P, Kantipong P, Jirajariyavej S, Sirivichayakul S, Munsakul W, Prasithsirikul W, Sungkanuparph S, Bowonwattanuwong C, Klinbuayaem V, Petoumenos K, Hirschel B, Bhakeecheep S, Ruxrungtham K. Etravirine and rilpivirine resistance in HIV-1 subtype CRF01_AE-infected adults failing non-nucleoside reverse transcriptase inhibitor-based regimens. Antivir Ther. 2011;16(7):1113-21. doi: 10.3851/IMP1906. PMID 22024527
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org